CLINICAL TRIAL: NCT01603888
Title: Molecular Forms of Plasma and Urinary B-type Natriuretic Peptide and Its N-terminal Prohormone in Health and Disease in Pediatric Cardiology
Status: Completed | Type: Observational
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Other Study IDs: bnp1-HMO-CTIL
Record Dates: First submitted 2012-05-20; First posted 2012-05-23 (Estimated); Last update posted 2017-11-28 (Actual); Status verified 2017-08

CONDITIONS: Heart Disease; Health
Keywords: children with heart disease; infants; healthy newborns
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional

GROUPS / COHORTS (3):
- healthy newborns, BNP, NT-proBNP: healthy newborns
  Interventions: Other: no intervention
- infants, BNP, NT-proBNP: infants
  Interventions: Other: no intervention
- children with heart disease, BNP, NT-proBNP: children with heart disease
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention

SUMMARY:
B-type natriuretic Peptide (BNP) is a cardiac hormone secreted from the cardiac myocytes in response to volume load. Plasma levels of BNP, as measured by immunoassay methods, are elevated in patients with heart diseases. However, the biological effects of BNP are blunted in heart failure and other cardiac conditions. Moreover, the peptide levels are also elevated in non cardiac conditions such as the neonatal period, sepsis and renal failure. Recent investigations suggest alteration of the peptide molecular structure in heart failure. These alterations may explain, at least partially, the reduced biological activities of BNP in heart failure.

Immunoreactive BNP and NT-proBNP have been identified in human urine. It has been suggested that urinary BNP correlates with plasma BNP, and may serve as a non-invasive measure for this cardiac marker. It is unclear what BNP fractions are cleared in the urine in health and disease.

The aim of the proposed studies is to elucidate precisely the molecular form of BNP in various disease and specific physiological states in plasma and urine of infants and children.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy newborn infants with normal pregnancy and delivery
2. Premature infants
3. Infants and children with heart disease who have NT-proBNP levels taken as part of cardiac evaluation

Exclusion Criteria:

1. Patients with non cardiac disease (renal, hepatic)
2. Patients with acute urinary disease or other acute non-cardiac diseases.

Max Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Normal newborn infants and premature babies. Infants and children with significant heart disease.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2013-01; Primary Completion 2015-01 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
molecular forms of BNP in healthy newborns, infants and children with heart disease. | one year
  Quantification of the specific molecular forms will be performed by liquid chromatography coupled to mass spectrometry.

SECONDARY OUTCOMES:
BNP presence and define its molecular forms in urine of healthy newborns,infants and children with heart disease. BNP presence and define its molecular forms in urine of healthy newborns and infant and children with heart disease. BNP presence and | one year
  Quantification of the specific molecular forms will be performed by liquid chromatography coupled to mass spectrometry.

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel